CLINICAL TRIAL: NCT04017923
Title: Age and Sex Related Changes in Nasal Tip Support
Brief Title: Measurement of Age and Sex Related Changes in Nasal Tip Support Using Digital Newton Meter
Status: Completed | Type: Observational
Sponsor: Baskent University Ankara Hospital (Other)
Responsible Party: Principal Investigator, Alper Koycu, Principal investigator, M.D., Baskent University Ankara Hospital
Other Study IDs: KA18/431
Record Dates: First submitted 2019-07-07; First posted 2019-07-12 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Nasal Valve Incompetence; Alar Collapse
Keywords: Nasal tip; Tip support; Rhinoplasty; Nasal cartilage; Age

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 20-29 age group
  Interventions: Diagnostic Test: measurement of nasal tip support in different age groups.
- 30-39 age group
  Interventions: Diagnostic Test: measurement of nasal tip support in different age groups.
- 40-64 age group
  Interventions: Diagnostic Test: measurement of nasal tip support in different age groups.
- 65 and older age group
  Interventions: Diagnostic Test: measurement of nasal tip support in different age groups.

INTERVENTIONS:
Diagnostic Test: measurement of nasal tip support in different age groups. — Nasal tip resistances , were measured in all age groups with a digital Newton meter.

SUMMARY:
Background:

It is predicted that the nasal tip support will decrease with aging due to weakening of cartilage and connective tissues. However, there is no consensus on the age at which this change began. It is quite difficult to evaluate the nasal tip support, while the ideal nasal tip support pressure is also not known. The aim of this study is to determine the nasal tip support pressure alterations in various age groups, by measuring nasal tip support with a Newton meter, according to age and gender.

Methods:

This prospective clinical study was conducted between January 2019 and April 2019 at a tertiary health facility. Nasal tip resistances in 4 different age groups, as 20-29, 30-39, 40-64 and 65 years and older, were measured with a digital Newton meter. A total number of 159 patients with a minimum of 36 patients in each age group were included in the study. Nasal tip resistance measurements were compared among nasal tip displacement distances of 2mm, 3mm and 4mm, according to age groups and gender.

ELIGIBILITY:
Inclusion Criteria:

* Four groups were formed as 20-29, 30-39, 40-64 and 65 years and older. A total of 159 patients with a minimum of 36 patients in each group were included in the study.

Exclusion Criteria:

* Patients with a history of nasal trauma, previous nasal surgery (septoplasty, rhinoplasty, tumor surgery), severe deviation of the caudal septum, visible external nasal deviation, and systemic disease affecting the connective tissue were excluded from the study.

Ages: 20 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Four groups were formed as 20-29, 30-39, 40-64 and 65 years and older
Sampling Method: Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Measurement of nasal tip resistance | All measurements were obtained within 2 months. (march 01-May 01)
  A digital newton meter was used to measure the nasal tip resistance

CONTACTS AND LOCATIONS:
Locations (1):
- Alper Koycu, Ankara, Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No